CLINICAL TRIAL: NCT04242927
Title: Efficacy of Nicotinic Acid for VEGFR Inhibitor-Associated Hand-Foot Skin Reactions in Solid Tumor Patients: a Randomised Controlled Phase 2 Trial
Brief Title: A Study to Investigate Nicotinic Acid on VEGFR Inhibitor-Associated Hand-Foot Skin Reactions
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: First People's Hospital of Hangzhou (Other)
Collaborators: Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: NAVI
Record Dates: First submitted 2020-01-23; First posted 2020-01-27 (Actual); Last update posted 2020-04-01 (Actual); Status verified 2020-03

CONDITIONS: Hand-Foot Skin Reaction (HFSR)
MeSH Terms: interventions — Niacin; Tablets

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Nicotinic acid + Routine care (Experimental): Nicotinic acid is administered orally at 50 mg (grade 2) or 100 mg (grade 3) three times daily with routine care.
  Interventions: Drug: Nicotinic acid +Routine care
- Routine care (Active Comparator): Routinely apply urea ointment and provide best supportive care.
  Interventions: Drug: Routine care

INTERVENTIONS:
Drug: Nicotinic acid +Routine care — Nicotinic acid is administered orally at 50 mg (grade 2) or 100 mg (grade 3) three times daily with routine care.
  Other Names: Nicotinic Acid 50 MG Oral Tablet
  Arms: Nicotinic acid + Routine care
Drug: Routine care — Routinely apply urea ointment and provide best supportive care.
  Other Names: Urea ointment
  Arms: Routine care

SUMMARY:
Hand-Foot Skin Reaction (HFSR) is a common adverse event induced by Vascular Endothelial Growth Receptor Inhibitor (VEGFRi) in cancer patients. The main purpose of this study is to evaluate the efficacy and safety of nicotinic acid in solid tumor patients with grade II/III VEGFRi-associated HFSR.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent obtained prior to performing any protocol-related procedures, including blood serum collecting
* HFSR grade 2 or higher after treatment with VEGFR inhibitors (such as sorafenib, regorafenib, anlotinib, and apatinib), according to NCI CTCAE V5.0 - PPE
* Age from 18 to 75 years.
* Life expectancy of at least 3 months at Day 1

Exclusion Criteria:

* History of allergy to B vitamins
* Major surgery or severe traumatic injury, fracture within 4 weeks prior to first dose of nicotinic acid or ulceration and any factors that significantly affect oral drug absorption, such as inability to swallow, chronic diarrhea, and intestinal obstruction
* Patient who takes isoniazid in combination with sorafenib and other VEGFR inhibitors.
* History of psychiatric drugs substance abuse and fails to quit it or has amental disorder
* Pregnant or nursing women, fertile patient who is unwilling or unable to use effective contraception

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2020-03-09 (Actual); Primary Completion 2021-03-09 (Estimated); Study Completion 2022-03-09 (Estimated)

PRIMARY OUTCOMES:
Response rate of VEGFR inhibitor-associated hand-foot skin reaction | 2 year
  Proportion of patients who achieve NCI CTCAE v5.0 - Palmar-Plantar Erythrodysesthesia (PPE) grade 0/1 (enrolled grade 2 patients) or grade 0-2 (enrolled grade 3 patients).
Complete response rate of VEGFR inhibitor-associated hand-foot skin reaction | 2 year
  Proportion of patients who achieve NCI CTCAE v5.0 - PPE grade 0.

SECONDARY OUTCOMES:
Dose adjustment/withdrawal ratio | 2 year
  Proportion of patients who need dose adjustment or withdrawal of VEGFR inhibitors, such as sorafenib, regorafenib, anlotinib, and apatinib.
Hand-Foot Reaction Quality of Life (HF-QoL) | 2 year
  Hand-Foot Reaction Quality of Life (HF-QoL) questionnaire, scoring results statistics. The HF-QoL symptom and daily activity total scores were transformed to a scale of 0 to 4, based on the sum of each unit-weighted item score divided by the maximum score. Higher scores on the HF-QoL indicate worse quality of life or greatersymptom burden.

CONTACTS AND LOCATIONS:
Overall Officials: Shenglin Ma, MD, Principal Investigator — First People's Hospital of Hangzhou
Locations (1):
- First People's Hospital of Hangzhou, Hangzhou, Zhejiang, China